CLINICAL TRIAL: NCT02843594
Title: A Study to Assess the Clinical Outcomes of Surgical Phaco Segmentation Techniques in Patients Undergoing Cataract Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iantech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEEP103
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- LEEP Intervention C1 (Active Comparator): Cataract surgery with micro-interventional LEEP technology lens fragmentation (non-randomized cohort 1)
  Interventions: Procedure: LEEP intervention
- LEEP Intervention C2 (Active Comparator): Cataract surgery with micro-interventional LEEP technology lens fragmentation (randomized cohort 2)
  Interventions: Procedure: LEEP intervention
- Control Phaco C2 (Placebo Comparator): Cataract surgery with conventional phaco-assisted lens fragmentation (randomized cohort 2)
  Interventions: Procedure: Standard Phaco Control

INTERVENTIONS:
Procedure: LEEP intervention — Low Energy Endosafe Phaco (LEEP) with micro-interventional lens fragmentation
  Arms: LEEP Intervention C1; LEEP Intervention C2
Procedure: Standard Phaco Control
  Arms: Control Phaco C2

SUMMARY:
The purpose of this research study is to evaluate the clinical outcomes of different cataract surgical techniques for lens fragmentation in subjects undergoing routine cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand study requirements, willing to follow study instructions and willing to return for required study follow-up visits as confirmed by provision of written informed consent.
2. Subjects with a visually significant cataract scheduled to undergo cataract surgery
3. Subjects > 18 years of age
4. BCVA at baseline not better than 20/40
5. Grade 1+ cataracts

Exclusion Criteria:

1. Subjects not able to complete the informed consent form
2. Subjects < 18 years of age
3. Polar cataracts
4. Zonular instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative Dispersed Phaco energy | Intraoperative
  Total phaco power and energy used as recorded by the phaco machine

SECONDARY OUTCOMES:
Endothelial cell loss | 1 month
  Change from baseline endothelial cell density as measured by specular microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica de Ojos Panama City, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ianchulev T, Chang DF, Koo E, MacDonald S, Calvo E, Tyson FT, Vasquez A, Ahmed IIK. Microinterventional endocapsular nucleus disassembly: novel technique and results of first-in-human randomised controlled study. Br J Ophthalmol. 2019 Feb;103(2):176-180. doi: 10.1136/bjophthalmol-2017-311766. Epub 2018 Apr 18. PMID 29669780